CLINICAL TRIAL: NCT06639646
Title: The Gut Brain Axis, Effect of Dietary Changes and Probiotics Supplement on Depression Symptoms
Brief Title: The Gut Brain Axis, Effect of Dietary Changes and Probiotics Supplement on Depression Symptoms .
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Salma Hosny Abd-allah Mohamed, Demonstrator in Family Medicine Department- Faculty of Medicine- Cairo University, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MD-257-2023
Record Dates: First submitted 2024-10-07; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Gut-brain Axis; Dietary Changes; Probiotics Supplement; Depression Symptoms
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary group (Experimental): A Dietary intervention group receiving health education message about healthy diet and probiotics supplements ( spores of poly antibiotic resistant "Lactobacilli 5 billion" in form of capsules registrated by the Egyption drug auyjority "EDA" and sold in Egyption markets under brand name "Lactèol Forte ®" capsules by Rameda® company.
  The probiotic supplement is recommended to be given twice daily for 12 wks duration.
  Interventions: Dietary Supplement: Probiotics supplements
- Control group (Active Comparator): A Control group receiving health education about healthy diet. At the end of the 12 wk. period, the same measurements are repeated.
  Interventions: Dietary Supplement: Health diet

INTERVENTIONS:
Dietary Supplement: Probiotics supplements — A Dietary intervention group receiving health education message about healthy diet and probiotics supplements ( spores of poly antibiotic resistant "Lactobacilli 5 billion" in form of capsules registrated by the Egyption drug auyjority "EDA" and sold in Egyption markets under brand name "Lactèol Forte ®" capsules by Rameda® company.
  The probiotic supplement is recommended to be given twice daily for 12 wks duration.
  Arms: Dietary group
Dietary Supplement: Health diet — A Control group receiving health education about healthy diet. At the end of the 12 wk. period, the same measurements are repeated
  Arms: Control group

SUMMARY:
To investigate the effects of a high-fiber diet and probiotic supplementation on depression symptoms in adult individuals.

DETAILED DESCRIPTION:
Depression is prevalent mental health disorder that significantly impacts individuals' quality of life. Despite the availability of effective treatments such as pharmacotherapy and psychotherapy, there are still significant limitations to these approaches. Medications can have unwanted side effects and may not be effective for all patients, while psychotherapy can be time-consuming and expensive. Furthermore, many individuals may not have access to these treatments due to financial, geographical, or cultural barriers.

A more recent study published in the Journal of Pediatric Gastroenterology and Nutrition in 2020 investigated the effects of a probiotic supplement on gastrointestinal symptoms and quality of life in children with functional abdominal pain. The study found that the probiotic supplement improved gastrointestinal symptoms and quality of life in the children.

Overall, while there is limited research on probiotics in Egypt, the available studies suggest that probiotics may have potential health benefits for various populations. However, further research is needed to better understand the optimal types, doses and duration of probiotic supplementation for specific health outcomes in Egyptian populations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals aged 18 to 65 years.
* Both sexes.

Exclusion Criteria:

* Pregnancy or lactation
* Recent use of antibiotics or corticosteroids (within the past 3 months)
* Chronic medical conditions that may interfere with study participation or interpretation of results (e.g., hypo or hyperthyroidism , cancer, diabetes, cardiovascular disease)
* Current or past diagnosis of major depressive disorder or anxiety disorder
* Current use of antidepressant or anxiolytic medications
* History of gastrointestinal disorders or diseases (e.g., inflammatory bowel disease, celiac disease , malabsorbtion )
* History of substance abuse or dependence

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Depression score using arabic version of PHQ9 | For 12 weeks after dietary supplement
  Depression score using arabic version of PHQ9 was recorded .The PHQ-9 (Patient Health Questionnaire-9) is a tool used to assess the severity of depression. It consists of nine questions, each related to symptoms experienced over the past two weeks. Each question is scored from 0 to 3, with the total score ranging from 0 to 27.

SECONDARY OUTCOMES:
The safety of the dietary | For 12 weeks after dietary supplement
  The safety of the dietary intervention and probiotics was recorded. Participants were asked to report any adverse events or intolerances related to the dietary changes or probiotic
Tolerability of the dietary intervention | For 12 weeks after dietary supplement
  Tolerability of the dietary intervention was recorded. Participants were asked to report any adverse events or intolerances related to the dietary changes or probiotic
Tolerability of probiotics | For 12 weeks after dietary supplement
  Tolerability of probiotics was recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data was available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data was available upon a reasonable request from the corresponding author.